CLINICAL TRIAL: NCT02941848
Title: A Randomized, Open-Label, Two-way Crossover, Single-Dose Study to Compare Pharmacokinetic Properties and Safety After Administration of HCP1306 Tablet and Co-administration of HGP0816 Tablet, HGP1404 Tablet in the Healthy Adults
Brief Title: Evaluate the Pharmacokinetics and Safety of HCP1306 and Co-administration of HGP0816, HGP1404 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROZE-102
Record Dates: First submitted 2016-10-11; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2015-01

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 (Experimental): C → A + B
  A : HGP0816 B : HGP1404 C : HCP1306
  Interventions: Drug: HGP0816; Drug: HGP1404; Drug: HCP1306
- Group2 (Experimental): A + B → C
  A : HGP0816 B : HGP1404 C : HCP1306
  Interventions: Drug: HGP0816; Drug: HGP1404; Drug: HCP1306

INTERVENTIONS:
Drug: HGP0816
Drug: HGP1404
Drug: HCP1306

SUMMARY:
The purpose of this study is to evaluate Pharmacokinetic Properties and Safety after administration of HCP1306 tablet and Co-administration of HGP0816 tablet, HGP1404 tablet in the healthy adults.

DETAILED DESCRIPTION:
A Randomized, Open-Label, Two-way Crossover, Single-Dose Study to Compare Pharmacokinetic Properties and Safety after administration of HCP1306 tablet and Co-administration of HGP0816 tablet, HGP1404 tablet in the healthy adults

ELIGIBILITY:
[Inclusion criteria]

1. Healthy adult of 19 to 50 of age at screening.
2. 18.5 ≤ Body mass index (BMI) < 25.

   ※ BMS (kg/m2)= body weight (kg)/[height (m)2]
3. Body weight ≥ 55 kg for men and ≥ 50 kg for women.
4. Individual considered by the responsible physician to be eligible as a subject based on the results of hematology test, blood chemistry test, immunoserology test, urinalysis, and electrocardiogram (ECG) as performed according to the characteristics of the drug (including those with not clinically significant (NCS) abnormalities).
5. Women must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and a negative pre-dose urine β-hCG test at a time point defined in the protocol and must be applicable to one of the followings.

   * Postmenopausal (no spontaneous menstruation for at least 2 years)
   * Surgical sterilization (sterilized by hysterectomy, bilateral ovariectomy or tubal ligation, or other methods)
   * A male partner is sterilized prior to screening (documented azoospermia following vasectomy) and this man is the subject's only partner.
   * The subject must agree to use adequate methods of contraception continuously and properly during the period of time from at least 14 days prior to the first dose to at least 28 days after the last dose of the investigational product.

     * Adequate methods of contraception include abstinence and physical barrier methods (e.g., condom, diaphragm, or cervical cap) and contraceptive devices or pills containing hormones that may have drug-drug interactions with the investigational product are not to be used during the study period, in principle.
6. Sexually active male subject with a female partner of childbearing potential must agree to avoid pregnancy (condom, etc.) during the study and to maintain adequate methods of contraception and not donate sperms during the study and for 28 days after the last dose of the investigational product (the methods of contraception are not necessary if the male subject or his female partner is sterile).
7. After receiving and understanding sufficient explanations about the study, the individual must voluntarily decide to participate in the study and provide written informed consent to complying with study instructions.

[Exclusion criteria]

1. Evidence or history of clinically significant diseases in the hepatobiliary system, kidney, nervous system, psychiatric system, respiratory system, endocrine system (thyroid dysfunction, etc.), hemato-oncology, cardiovascular system, immune system, or musculoskeletal system (myopathy, etc.).
2. History of gastrointestinal disorders (e.g., Crohn's disease, ulcerative colitis) or surgery (except for simple typhlotomy or hernia repair) that may affect the absorption of the investigational product.
3. Hypersensitivity reactions to any of the components of the investigational product or its excipients or drugs of the same class.
4. Hereditary disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
5. Vital signs measured in the sitting position after at least 5 minutes of rest as follows: systolic blood pressure (SBP) > 150 mmHg or < 90 mmHg or diastolic blood pressure (DBP) > 100 mmHg or < 50 mmHg.
6. Screening clinical laboratory test results as follows:

   * Blood total bilirubin level > 1.5 x upper limit of normal (ULN)
   * Blood aspartate aminotransferase (AST, also known as serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT, also known as serum glutamate pyruvate transaminase [SGPT]) > 1.25 x ULN
   * Blood urea nitrogen (BUN) > 25.0 mg/dL or creatinine > 1.4 mg/dL
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation

     ※ eGFR (mL/min/1.73m2) = 175 x [serum creatinine (mg/dL)]-1.154 x [age (years)]-0.203 (X 0.742, if female)
   * Blood Creatinine Phosphokinase (CK) > 2 x ULN
7. History of significant drug abuse within 1 year of screening or positive urine drug test results.
8. Administration of drugs within 30 days of the investigational product administration that are expected to or may affect the metabolism of the investigational product.
9. Administration of the following drugs within the relevant period, except for local agents without significant systemic absorption and hormonal contraceptives.

   * Ethical (ETC) drugs within 14 days of the first investigational product administration
   * Over-the-counter (OTC) drugs including health foods and vitamin preparations within 7 days of the first investigational product administration
   * Drugs administered via depot injection or other implantations (except for contraceptives) within 30 days of the first investigational product administration
10. Significant alcohol dependency within 1 year of screening, continuous drinking within 6 months of screening (> 210 g/week), or unable to refrain from drinking during the study period starting from 2 days prior to the first investigational product administration.
11. Continuous caffeine intake (e.g., coffee > 5 cups/day, tea > 1250 cc/day, cola > 1250 cc/day) or unable to refrain from caffeine intake during the study period starting from 2 days prior to the first investigational product administration.
12. Continuous smoking (> 10 cigarettes/day) or unable to refrain from smoking during the study period starting from 2 days prior to the first investigational product administration.
13. Intake of grapefruits or foods containing grapefruits within 7 days prior to the first investigational product administration.
14. Participation in another clinical trial (including a bioequivalence study) and administration of another investigational product within 60 days prior to the investigational product administration in this study (3 months for biologics; a prolonged period of time may be applied with half life taken into account).
15. Whole blood donation within 60 days or apheresis donation within 30 days prior to the investigational product administration.
16. Pregnant or lactating women.
17. Subject considered by the investigator to be inappropriate for study participation due to other reasons.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
AUClast of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
Cmax of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
AUClast of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
Cmax of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours

SECONDARY OUTCOMES:
AUCinf of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
tmax of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
t1/2 of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
CL/F of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
Vd/F of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
MRT of Rosuvastatin | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
AUCinf of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
Tmax of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
T1/2 of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
CL/F of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
Vd/F of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours
MRT of Free Ezetimibe | Pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Choon Ok Kim, MD, Principal Investigator — Yonsei University Health System, Severance Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Min KL, Park MS, Jung J, Chang MJ, Kim CO. Comparison of Pharmacokinetics and Safety of a Fixed-dose Combination of Rosuvastatin and Ezetimibe Versus Separate Tablets in Healthy Subjects. Clin Ther. 2017 Sep;39(9):1799-1810. doi: 10.1016/j.clinthera.2017.07.038. Epub 2017 Aug 10. PMID 28803122